CLINICAL TRIAL: NCT03683732
Title: EXTENSION OF THE EUROPEAN E-BUG PROJECT TOWARDS 15-18 YEARS - How to Raise Awareness About Antibiotics and Vaccination Among Frenchteenagers -
Brief Title: EXTENSION OF THE EUROPEAN E-BUG PROJECT
Acronym: Ext EBUG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 18-DSP-02
Record Dates: First submitted 2018-09-17; First posted 2018-09-25 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Vaccination Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Frenchteenagers
  Interventions: Behavioral: Individual semi-structured interviews

INTERVENTIONS:
Behavioral: Individual semi-structured interviews — Individual semi-structured interviews were conducted using purposeful sampling of 15- to 18-year-olds, until data saturation, and were transcribed and analysed

SUMMARY:
Bacterial resistance to antibiotics is a growing concern in Europe, vaccination coverage is inadequate, and young adults, who are the highest antibiotic consumers, have the lowest level of knowledge. Extension of the e-Bug project, a European educational school programme concerning microbes, antibiotics and vaccination, to 15-18-year-olds implies the development of educational resources based on social marketing to promote sustainable behavioural changes. The objectives of the present study, which is part of the needs assessment in France, are to explore the attitudes, knowledge and behaviour of 15-18-year-olds concerning antibiotics and vaccination and their health education needs.

Individual semi-structured interviews were conducted using purposeful sampling of 15- to 18-year-olds, until data saturation, and were transcribed and analysed.

ELIGIBILITY:
Inclusion Criteria:

* 15-18 year olds, various origines, studying in various pathways of higher secondary education or working.

Exclusion Criteria:

-

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The recrutement and the conversations were realized on a voluntary basis in the crossroads health young people of Nice, structure dedicated to the grown-up young adolescentset from 12 to 25 years old.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2013-12-05 (Actual)

PRIMARY OUTCOMES:
Behavior concerning antibiotics and vaccination | 5 years
  questionnary (no scale) used to Explore attitudes, behavior and knowledge of the 15-18-year-old young people in France concerning antibiotics and vaccination . Data collection by means of a questionnary during a unique interview with the teenager.

SECONDARY OUTCOMES:
Expectation and media | 5 years
  questionnary (no scale) used to Determine the expectations of the 15-18-year-old young people in France and needs concerning the methods and the supports of education. Data collection by means of a questionnary during a unique interview with the teenager

CONTACTS AND LOCATIONS:
Overall Officials: Pia Touboul, Dr, Study Chair — Centre Hospitalier Universitaire de Nice